CLINICAL TRIAL: NCT00716820
Title: Outcome Survey Of Specific Use Of 12.5 Mg Sutent Capsule Against Gastrointestinal Stromal Tumor: Implementation Guidelines.
Brief Title: Special Investigation For Gist Of Sunitinib Malate (Regulatory Post Marketing Commitment Plan).
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181175
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SUNITINIB MALATE: Patients taking Sutent.
  Interventions: Drug: SUNITINIB MALATE

INTERVENTIONS:
Drug: SUNITINIB MALATE — SUTENT capsule 12.5 mg, depending on the Investigator prescription. Frequency and duration are according to Package Insert as follows. "The usual adult dosage for oral sunitinib is 50 mg once daily, 4 weeks on followed by 2 weeks off (Schedule 4/2). This comprises 1 treatment cycle, which may be repeated.
  The dosage may be decreased according to the patient's clinical condition."
  Other Names: SUTENT

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first SUNITINIB MALATE(Sutent) should be registered.

ELIGIBILITY:
Inclusion Criteria:

Patients need to be administered SUNITINIB MALATE(Sutent) in order to be enrolled in the surveillance.

Exclusion Criteria:

Patients not administered SUNITINIB MALATE(Sutent).

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A6181175 prescribes the SUNITINIB MALATE(Sutent).
Sampling Method: Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181175&StudyName=Special%20Investigation%20For%20Gist%20Of%20Sunitinib%20Malate%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib Malate: Usually, 50 mg of sunitinib malate was orally administered to adult participants once daily in repetitive cycles of 4 weeks on treatment followed by 2 weeks off according to Japanese package insert.
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 472
Completed | 472
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 472
Age, Customized [Number; unit: Participants]
  <15 years | 0
  >=15 and <65 years | 238
  ˃=65 years | 227
  Unknown | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175
  Male | 297

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 2 Years
Population: Safety analysis set comprised of participants who had met the inclusion criteria and had received sunitinib malate at least once.
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 472
Participants | 450

2. Primary Outcome: Objective Response Rate
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). The result was presented along with the corresponding exact 2-sided 95% confidence interval (CI).
Time Frame: MAX 2 Years
Population: Efficacy analysis set comprised of participants in safety analysis set who had efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 389
Percentage of participants | 20.1 [16.2 to 24.4]

3. Secondary Outcome: Objective Response Rates by KIT Expression Status
Description: Percentage of participants with objective response based assessment of CR or confirmed PR according to RECIST. Objective response rates by KIT expression status were calculated according to RECIST and were presented along with the corresponding exact 2-sided 95% CIs.
Time Frame: MAX 2 Years
Population: Efficacy analysis set comprised of participants in safety analysis set who had efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- KIT Positive: Participants with positive KIT expression who received sunitinib malate according to Japanese package insert
- KIT Negative: Participants with negative KIT expression who received sunitinib malate according to Japanese package insert
- Unknown: Participants with unknown KIT expression status who received sunitinib malate according to Japanese package insert
Arm/Group | KIT Positive | KIT Negative | Unknown
Number analyzed (Participants) | 339 | 8 | 42
Percentage of participants | 21.2 [17.0 to 26.0] | 12.5 [0.3 to 52.7] | 11.9 [4.0 to 25.6]

4. Secondary Outcome: Objective Response Rates by c-Kit Mutation Status
Description: Percentage of participants with objective response based assessment of CR or confirmed PR according to RECIST. Objective response rates by c-kit mutation status were calculated according to RECIST and were presented along with the corresponding exact 2-sided 95% CIs.
Time Frame: MAX 2 Years
Population: Efficacy analysis set comprised of participants in safety analysis set who had efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- c-Kit With Mutation: Participants with c-kit mutation who received sunitinib malate according to Japanese package insert
- c-Kit Without Mutation: Participants without c-kit mutation who received sunitinib malate according to Japanese package insert
- Unknown: Participants with unknown c-kit mutation status who received sunitinib malate according to Japanese package insert
Arm/Group | c-Kit With Mutation | c-Kit Without Mutation | Unknown
Number analyzed (Participants) | 77 | 15 | 297
Percentage of participants | 22.1 [13.4 to 33.0] | 20.0 [4.3 to 48.1] | 19.5 [15.2 to 24.5]

5. Secondary Outcome: Objective Response Rates by Platelet - Derived Growth Factor Receptor Alpha (PDGFRα) Mutation Status
Description: Percentage of participants with objective response based assessment of CR or confirmed PR according to RECIST. Objective response rates by PDGFRα mutation status were calculated according to RECIST and were presented along with the corresponding exact 2-sided 95% CIs.
Time Frame: MAX 2 Years
Population: Efficacy analysis set comprised of participants in safety analysis set who had efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PDGFRα With Mutation: Participants with PDGFRα mutation who received sunitinib malate according to Japanese package insert
- PDGFRα Without Mutation: Participants without PDGFRα mutation who received sunitinib malate according to Japanese package insert
- Unknown: Participants with unknown PDGFRα mutation status who received sunitinib malate according to Japanese package insert
Arm/Group | PDGFRα With Mutation | PDGFRα Without Mutation | Unknown
Number analyzed (Participants) | 5 | 36 | 348
Percentage of participants | 20.0 [0.5 to 71.6] | 27.8 [14.2 to 45.2] | 19.3 [15.2 to 23.8]

6. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events in Elderly Population
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). Elderly population was defined as the participants who aged 65 or older.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Elderly: Participants aged ˃=65 years who received sunitinib malate according to Japanese package insert
- Non-elderly: Participants aged ˂65 years who received sunitinib malate according to Japanese package insert
- Unknown: Participants with unknown age who received sunitinib malate according to Japanese package insert
Arm/Group | Elderly | Non-elderly | Unknown
Number analyzed (Participants) | 227 | 238 | 7
Participants | 220 | 226 | 4

7. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Who Had Hepatic Impairment
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). Hepatic impairment referred not to transient laboratory test value abnormalities, but to the events that were clinically noteworthy and required follow-up.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With Hepatic Impairment: Participants with baseline hepatic impairment who received sunitinib malate according to Japanese package insert
- Without Hepatic Impairment: Participants without baseline hepatic impairment who received sunitinib malate according to Japanese package insert
- Unknown: Participants with no information on baseline hepatic impairment who received sunitinib malate according to Japanese package insert
Arm/Group | With Hepatic Impairment | Without Hepatic Impairment | Unknown
Number analyzed (Participants) | 55 | 412 | 5
Participants | 52 | 394 | 4

8. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Who Had Renal Impairment
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). Renal impairment referred not to transient laboratory test value abnormalities, but to the events that were clinically noteworthy and required follow-up.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With Renal Impairment: Participants with baseline renal impairment who received sunitinib malate according to Japanese package insert
- Without Renal Impairment: Participants without baseline renal impairment who received sunitinib malate according to Japanese package insert
- Unknown: Participants with no information on baseline renal impairment who received sunitinib malate according to Japanese package insert
Arm/Group | With Renal Impairment | Without Renal Impairment | Unknown
Number analyzed (Participants) | 52 | 416 | 4
Participants | 47 | 400 | 3

9. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Who Used Concomitant Cytochrome P450 3A4 (CYP3A4) Inhibitors
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). A total of 38 drugs including tofisopam, bromocriptin mesilate, and fluvoxamine maleate were defined as CYP3A4 inhibitors.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With Concomitant CYP3A4 Inhibitors (Start of Treatment): Participants with concomitant CYP3A4 inhibitors at start of sunitinib malate treatment according to Japanese package insert
- With Concomitant CYP3A4 Inhibitors (During Treatment): Participants with concomitant CYP3A4 inhibitors during sunitinib malate treatment according to Japanese package insert
- Without Concomitant CYP3A4 Inhibitors: Participants without concomitant CYP3A4 inhibitors on sunitinib malate treatment according to Japanese package insert
Arm/Group | With Concomitant CYP3A4 Inhibitors (Start of Treatment) | With Concomitant CYP3A4 Inhibitors (During Treatment) | Without Concomitant CYP3A4 Inhibitors
Number analyzed (Participants) | 12 | 12 | 448
Participants | 12 | 12 | 426

10. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events Who Were Under Long-Term Treatment
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). The long-term treatment was defined as the treatment continued more than 24 weeks.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 472
Participants | 3

11. Secondary Outcome: Numbers of Participants With Treatment-Related Adverse Events Corresponded to Items for Priority Investigation
Description: The following adverse events were defined as items for priority investigation : (1) lung disorder including interstitial pneumonia, (2) bone marrow depression including platelets decreased, white blood cell decreased, and anaemia, (3) haemorrhage including those due to tumor degeneration or shrinkage, (4) cardiac function disturbance including QT interval prolonged and left ventricular ejection fraction decreased, (5) dysfunction adrenal, (6) pancreatic dysfunction including lipase increased, (7) thyroid function decreased, (8) cutaneous symptoms (hand and foot syndrome), (9) serious infections, (10) rhabdomyolysis, myopathy, and (11) reversible posterior leukoencephalopathy syndrome (RPLS). Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 472
Participants
  Lung disorder | 1
  Bone marrow depression | 386
  Haemorrhage | 106
  Cardiac function disturbance | 29
  Dysfunction adrenal | 1
  Pancreatic dysfunction | 53
  Thyroid function decreased | 142
  Cutaneous symptoms (hand and foot syndrome) | 223
  Serious infections | 20
  Rhabdomyolysis, myopathy | 17
  RPLS | 4

12. Other Pre Specified Outcome: Number of Participants With Treatment-Related Serious Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. A treatmen-trelated serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 472
Participants | 201

13. Other Pre Specified Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 472
Participants | 98

14. Other Pre Specified Outcome: Number of Participants With Treatment-Related Adverse Events Grade 3 or Higher in Common Toxicity Criteria for Adverse Events (CTCAE)
Description: A treatment-related adverse event was any untoward medical occurrence attributed to sunitinib malate in a participant who received sunitinib malate. Relatedness to sunitinib malate was assessed by the investigator and sponsor (Pfizer Japan Inc.). The severity for each adverse event was assessed according to CTCAE as follows: grade 3, severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, or disabling; grade 4, life-threatening consequences or urgent intervention indicated; grade 5, death related to adverse event.
Time Frame: MAX 2 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 472
Participants | 334

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 259/472
Other Adverse Events (participants affected / at risk) | 429/472
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate (N=472)
Pneumonia staphylococcal (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Cholangitis infective (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Neutropenic infection (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Gingival abscess (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Abscess (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Abdominal abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hypopituitarism (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Aneurysm (Vascular disorders) | 1
Aneurysm ruptured (Vascular disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Enterocolonic fistula (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatic enzyme abnormality (Gastrointestinal disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Vesical fistula (Renal and urinary disorders) | 1
Face oedema (General disorders) | 1
Pain (General disorders) | 1
Amylase increased (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 1
Protein urine present (Investigations) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Septic shock (Infections and infestations) | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hyperammonaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Melaena (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 2
Cholangitis acute (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 2
Renal disorder (Renal and urinary disorders) | 2
Multi-organ failure (General disorders) | 2
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 2
Red blood cell count decreased (Investigations) | 2
Bone marrow failure (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 3
Hepatic encephalopathy (Nervous system disorders) | 3
Cardiac failure (Cardiac disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Liver disorder (Hepatobiliary disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 3
Blood creatine phosphokinase increased (Investigations) | 3
Sepsis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Dehydration (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Ileus (Gastrointestinal disorders) | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 4
Malaise (General disorders) | 4
Death (General disorders) | 4
Fatigue (General disorders) | 4
Blood creatinine increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 5
Infection (Infections and infestations) | 6
Haemorrhage (Vascular disorders) | 6
Aspartate aminotransferase increased (Investigations) | 6
Haemoglobin decreased (Investigations) | 6
Hepatic function abnormal (Hepatobiliary disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 8
Hypothyroidism (Endocrine disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Hypertension (Vascular disorders) | 11
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 12
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13
Decreased appetite (Metabolism and nutrition disorders) | 15
Pyrexia (General disorders) | 19
Anaemia (Blood and lymphatic system disorders) | 26
Neutrophil count decreased (Investigations) | 33
Disease progression (General disorders) | 41
White blood cell count decreased (Investigations) | 41
Platelet count decreased (Investigations) | 90
Nausea (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Alanine aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 5
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate (N=472)
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Neutropenia (Blood and lymphatic system disorders) | 10
Bone marrow failure (Blood and lymphatic system disorders) | 7
Leukopenia (Blood and lymphatic system disorders) | 10
Anaemia (Blood and lymphatic system disorders) | 61
Left ventricular dysfunction (Cardiac disorders) | 6
Hypothyroidism (Endocrine disorders) | 113
Hyperthyroidism (Endocrine disorders) | 17
Eyelid oedema (Eye disorders) | 5
Nausea (Gastrointestinal disorders) | 68
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 96
Cheilitis (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 116
Haemorrhoids (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 12
Abdominal pain upper (Gastrointestinal disorders) | 7
Glossitis (Gastrointestinal disorders) | 7
Ascites (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 28
Abdominal discomfort (Gastrointestinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 34
Vomiting (Gastrointestinal disorders) | 46
Proctalgia (Gastrointestinal disorders) | 5
Anal haemorrhage (Gastrointestinal disorders) | 5
Pancreatic enzyme abnormality (Gastrointestinal disorders) | 6
Performance status decreased (General disorders) | 7
Face oedema (General disorders) | 15
Chest pain (General disorders) | 8
Malaise (General disorders) | 58
Mucosal inflammation (General disorders) | 7
Pyrexia (General disorders) | 67
Fatigue (General disorders) | 56
Oedema (General disorders) | 43
Oedema peripheral (General disorders) | 20
Hepatic function abnormal (Hepatobiliary disorders) | 21
Liver disorder (Hepatobiliary disorders) | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 9
Periodontitis (Infections and infestations) | 6
Gingivitis (Infections and infestations) | 24
Nasopharyngitis (Infections and infestations) | 15
C-reactive protein increased (Investigations) | 9
Gamma-glutamyltransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 40
Amylase increased (Investigations) | 19
Alanine aminotransferase increased (Investigations) | 24
Haematocrit decreased (Investigations) | 5
Haemoglobin decreased (Investigations) | 65
Lipase increased (Investigations) | 17
Lymphocyte count decreased (Investigations) | 13
Ejection fraction decreased (Investigations) | 11
Blood pressure increased (Investigations) | 6
Platelet count decreased (Investigations) | 216
Blood alkaline phosphatase increased (Investigations) | 16
Blood albumin decreased (Investigations) | 11
Blood creatinine increased (Investigations) | 26
Blood creatine phosphokinase increased (Investigations) | 14
Blood bilirubin increased (Investigations) | 25
Blood thyroid stimulating hormone increased (Investigations) | 27
Blood uric acid increased (Investigations) | 8
Blood urea increased (Investigations) | 10
Neutrophil count decreased (Investigations) | 115
Red blood cell count decreased (Investigations) | 11
Weight decreased (Investigations) | 6
White blood cell count decreased (Investigations) | 188
Hyperamylasaemia (Metabolism and nutrition disorders) | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 10
Hyperlipasaemia (Metabolism and nutrition disorders) | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 10
Decreased appetite (Metabolism and nutrition disorders) | 101
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15
Hypokalaemia (Metabolism and nutrition disorders) | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 15
Hypoaesthesia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 27
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 49
Insomnia (Psychiatric disorders) | 14
Renal impairment (Renal and urinary disorders) | 10
Proteinuria (Renal and urinary disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 34
Pruritus (Skin and subcutaneous tissue disorders) | 13
Yellow skin (Skin and subcutaneous tissue disorders) | 22
Erythema (Skin and subcutaneous tissue disorders) | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 209
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 40
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 12
Dermatitis (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 6
Skin disorder (Skin and subcutaneous tissue disorders) | 9
Skin discolouration (Skin and subcutaneous tissue disorders) | 25
Hypertension (Vascular disorders) | 163
Haemorrhage (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.